CLINICAL TRIAL: NCT02484859
Title: Comparison of Normotensive Anesthesia Using a Combination of Metoprolol and Tramadol With Controlled Hypotension Using Remifentanil in Endoscopic Sinus Surgery
Brief Title: Comparison of Metoprolol and Tramadol With Remifentanil in Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Başar Erdivanlı, Asst. Prof., Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2015/14
Record Dates: First submitted 2015-06-19; First posted 2015-06-30 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Nasal Polyps
Keywords: Drug: remifentanil; Drug: tramadol; Drug: metoprolol; Functional endoscopic sinus surgery; Controlled hypotension
MeSH Terms: conditions — Nasal Polyps | interventions — Remifentanil; Tramadol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- remifentanil (Active Comparator): Following an intravenous bolus dose of 0.5 µg/kg remifentanil administered just before the induction of anaesthesia, patients will receive an intravenous infusion of remifentanil at a dose of 0.25-0.5 µg/kg/min throughout the surgery. The rate of infusion will be adjusted to maintain a mean blood pressure within %70-80 of the baseline value. At the end of the surgery, the rate of infusion will be decreased to 0.05 µg/kg/min, and continued until the patient is extubated.
  Interventions: Drug: Remifentanil
- tramadol + metoprolol (Active Comparator): Just before the induction of anaesthesia, an intravenous infusion of 1 mg/kg of tramadol in 100 ml isotonic fluid will be started. The infusion will be completed in 30 minutes using a perfusor. Additionally, following the administration of the neuromuscular blocking agent, 0.1 mg/kg of intravenous metoprolol will be administered within 5 minutes.
  Interventions: Drug: Tramadol; Drug: Metoprolol

INTERVENTIONS:
Drug: Remifentanil — Remifentanil infusion will be started with a bolus dose of 0.5 µg/kg before the induction, and will be continued throughout the surgery at a dose of 0.25-0.5 µg/kg/min. At the end of the surgery, the rate of infusion will be decreased to 0.05 µg/kg/min, and continued until the patient is extubated.
  Other Names: Ultiva
  Arms: remifentanil
Drug: Tramadol — 1 mg/kg tramadol will be added to 100 ml of isotonic fluid, and will be administered intravenously in exactly 30 minutes via a perfusor. The infusion will be started just before the induction.
  Other Names: Contramal
  Arms: tramadol + metoprolol
Drug: Metoprolol — 0.1 mg/kg of metoprolol will be administered intravenously within 5 minutes following the administration of neuromuscular blocking agent.
  Other Names: Beloc
  Arms: tramadol + metoprolol

SUMMARY:
Functional endoscopic sinus surgery (FESS) is indicated in diseases such as chronic sinusitis refractory to medical treatment, nasal polyposis, mass lesions in the nasal cavity. The purpose of this study is to determine whether tramadol and metoprolol are as effective as remifentanil in providing controlled hypotension during FESS.

DETAILED DESCRIPTION:
This study aims to compare two techniques for controlled hypotension during FESS. In both cases, the patients will be evaluated during the preoperative anesthetic visit, and will be given care by an anesthesiologist during the perioperative period.

Patients who are scheduled for an elective FESS operation will be included in the study. During the preoperative anaesthetic visit, patients who do not meet any of the the exclusion criteria will be offered to participate in hte study. Patients accepting to contribute tot he study will be randomised into one of the two groups via closed envelope technique.

A pilot study with 20 patients resulted in similar means and slightly different standard deviations of mean blood pressure. This pilot study showed that 44 patients in each group are sufficient to obtain 80% power with an alpha error of 0.05 and beta error of 20%. To compensate for missing/inconsistent data, or allow for better matching of the demographic variables, 3-5 additional patients will be recruited.

The anesthesiologist in charge of the patient will not be blinded to the groups, and will be responsible for maintaining the hypotension (and patient safety) with either remifentanil in one group, or tramadol and metoprolol in the other group. Systolic, diastolic, and mean blood pressures, and heart rate will be recorded into a spreadsheet every three minutes during the anaesthetic and surgical period. The data will be recorded via an excel form, which will validate the entries upon entrance. The accuracy and completeness of registry data will be verified by a third investigator, who will compare the registry data to the medical monitor records at the end of each operative day.

The surgeon will be blinded to the groups, and will be responsible for scoring the surgical vision and bleeding with the intraoperative bleeding score. The study drugs will be administered via the same type of infusion pump to facilitate the blinding process.

Any adverse event will be reported in the patient chart and study records.

Statistical analysis will be carried out using R and Statistical Package for the Social Sciences (SPSS) programs. Demographic variables (age, gender, American Society of Anesthesiologists (ASA) score, comorbidities) will be analysed using descriptive statistics. Study variables such as duration of operation, variance of the hemodynamic parameters, amount of bleeding, bleeding score, occurrence of adverse events will be analysed with the appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of rhinosinusitis
* indication for functional endoscopic sinus surgery

Exclusion Criteria:

* American Society of Anesthesiologists risk score > 2
* undertreated hypertension
* Haemoglobin A1c test level > 7.5
* pregnancy
* concurrent surgery
* history of drug abuse
* history of or new diagnosis of allergy to any of the study drugs
* history of post-operative nausea and vomiting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Başar Erdivanlı, Asst. Prof., Principal Investigator — Recep Tayyip Erdogan University, Medical Faculty, Department of Anesthesiology
Locations (1):
- Recep Tayyip Erdogan University, Rize, Eastern Blacksea, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We are still evaluating the guideline of the Medical Research Council (MRC) Hubs for Trials Methodology Research (HTMR) for individual participant data sharing.

REFERENCES:
- [Background] Hosemann W, Draf C. Danger points, complications and medico-legal aspects in endoscopic sinus surgery. GMS Curr Top Otorhinolaryngol Head Neck Surg. 2013 Dec 13;12:Doc06. doi: 10.3205/cto000098. PMID 24403974
- [Background] Cincikas D, Ivaskevicius J, Martinkenas JL, Balseris S. A role of anesthesiologist in reducing surgical bleeding in endoscopic sinus surgery. Medicina (Kaunas). 2010;46(11):730-4. PMID 21467830
- [Background] Lin D, Dalgorf D, Witterick IJ. Predictors of unexpected hospital admissions after outpatient endoscopic sinus surgery: retrospective review. J Otolaryngol Head Neck Surg. 2008 Jun;37(3):309-11. PMID 19128632
- [Background] Komatsu R, Turan AM, Orhan-Sungur M, McGuire J, Radke OC, Apfel CC. Remifentanil for general anaesthesia: a systematic review. Anaesthesia. 2007 Dec;62(12):1266-80. doi: 10.1111/j.1365-2044.2007.05221.x. PMID 17991265
- [Background] Rathjen T, Bockmuhl U, Greim CA. [Modern anesthesiologic concepts supporting paranasal sinus surgery]. Laryngorhinootologie. 2006 Jan;85(1):20-3. doi: 10.1055/s-2005-870562. German. PMID 16444651
- [Background] Khalil HS, Nunez DA. Functional endoscopic sinus surgery for chronic rhinosinusitis. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004458. doi: 10.1002/14651858.CD004458.pub2. PMID 16856048
- [Background] Sartcaoglu F, Celiker V, Basgul E, Yapakci O, Aypar U. The effect of hypotensive anaesthesia on cognitive functions and recovery at endoscopic sinus surgery. Eur J Anaesthesiol. 2005 Feb;22(2):157-9. doi: 10.1017/s0265021505230284. No abstract available. PMID 15816598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period started at 27.06.2015. Recruitment was performed by an anaesthesiologist at the outpatient polyclinic for anaesthesiology.
Pre-assignment Details: A total of 105 patients were evaluated. Three patients declined to participate in the study. Eleven patients did not meet inclusion criteria. On 29 December 2015, we reached the target number of patients (88). Since patients were matched for severity of sinonasal disease, we evaluated three more patients anticipating possible dropouts.
Period: Overall Study
Arm/Group | Remifentanil | Tramadol + Metoprolol
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil | Tramadol + Metoprolol | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (10.1) | 39.3 (10.6) | 38.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 28 | 32 | 60
American Society of Anesthesiologists physical status [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) physical status 1 denotes a normal healthy patient. This means a healthy, non-smoking person who exhibits no or minimal alcohol use.
  ASA physical status 2 denotes a patient with mild systemic disease (mild diseases only without substantive functional limitations). Examples include (but not limited to): current smoker, social alcohol drinker, pregnancy, obesity (30 < body mass index < 40), well-controlled diabetes mellitus/hypertension, mild lung disease.
  Participants
    1 | 24 | 25 | 49
    2 | 20 | 19 | 39
Lund-Mackay score [Median (Inter-Quartile Range); unit: units on a scale] — Various staging systems have been proposed for use in chronic rhinosinusitis. Many studies use the Lund-Mackay scale to evaluate radiographic images. This scale grades the right and left sides independently, looking at the maxillary, anterior ethmoids, posterior ethmoids, sphenoid, and frontal sinuses, as well as the ostiomeatal complex. Each sinus is scored a 0 (no abnormality), 1 (partial opacification), or 2 (total opacification), while the ostiomeatal complex is scored either a 0 or 2 (for presence or absence of disease). Scores range from 0-24.
  units on a scale | 12 [8.75 to 15] | 10 [6 to 14] | 11 [7 to 14.25]
Prothrombin time [Mean (Standard Deviation); unit: seconds] — Prothrombin time is a blood test that measures the time it takes for the liquid portion of the blood to clot. If a person is not taking blood thinning medicines, the normal range is 11 to 13.5 seconds.
  seconds | 13.1 (0.5) | 13.4 (0.6) | 13.3 (0.6)
Partial thromboplastin time [Mean (Standard Deviation); unit: seconds] — Partial thromboplastin time is a blood test that looks at how long it takes for blood to clot. In general, clotting should occur within 25 to 35 seconds. If the person is taking blood thinners, clotting takes up to two-and-a-half times longer.
  seconds | 30.6 (2.2) | 29.7 (2.2) | 30.1 (2.3)
International normalized ratio [Mean (Standard Deviation); unit: international normalized ratio] — Prothrombin time is a blood test that measures the time it takes for the liquid portion (plasma) of the blood to clot. Prothrombin time is measured in seconds. Most of the time, results are given as what is called international normalized ratio (INR).
  international normalized ratio | 1.01 (0.07) | 1.02 (0.08) | 1.01 (0.07)
Haemoglobin [Mean (Standard Deviation); unit: grams per deciliter] — The haemoglobin test is a blood test that measures how much haemoglobin is in the blood. Haemoglobin is a protein in red blood cells that carries oxygen. Normal results for adults vary, but in general are:
  Male: 13.8 to 17.2 grams per deciliter (g/dl) Female: 12.1 to 15.1 g/dl
  grams per deciliter | 14.1 (1.3) | 14.2 (1.3) | 14.2 (1.3)
Platelet count [Mean (Standard Deviation); unit: 10^3 platelets per microliter] — A platelet count is a lab test to measure how many platelets are present in the blood. Platelets are parts of the blood that help the blood clot. The normal number of platelets in the blood is 150 000 to 400 000 platelets per microliter (mcl). Normal value ranges may vary slightly.
  10^3 platelets per microliter | 236 (69) | 242 (69) | 239 (69)

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Bleeding Score
Description: Intraoperative bleeding score is reported by the surgeon according to Boezaart Surgical Field Grading scale. The scale ranges from 0 to 5. '0' is the best, and '5' is the worst outcome.
  The scale construct is:
  0 No bleeding.
  1. Slight bleeding, no suction is required.
  2. Slight bleeding, occasional suctioning required.
  3. Slight bleeding, frequent suctioning required. Bleeding threatens surgical field a few seconds after suction is removed.
  4. Moderate bleeding, frequent suctioning required. Bleeding threatens surgical field as soon as suction is removed.
  5. Severe bleeding, constant suctioning required. Bleeding appears faster than suctioning.
  Thoroughout the intraoperative period, the surgeon is free to report a score at any time he/she sees appropriate.
Time Frame: throughout surgery, up to 3 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remifentanil | Tramadol + Metoprolol
Number analyzed (Participants) | 44 | 44
units on a scale | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: Remifentanil vs Tramadol + Metoprolol; Median intraoperative bleeding scores were compared with Wilcoxon test. In this pilot study the power analysis showed that a sample size of 44 patients in each group was sufficient to detect a difference of 0.2 in the mean (standard deviation of 0.4) with an 80% power with an alpha error of 0.05 and a beta error of 20%. The Shapiro-Wilk test was used to test the distribution of data; Test type: Superiority; p > 0.69, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to Achieve Intraoperative Bleeding Score < 3
Description: The intraoperative bleeding score will be reported by the surgeon throughout surgery. At the start of the surgery, a timer will be used to measure the duration to achieve a bleeding score of 2.
Time Frame: throughout surgery, up to 20 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Remifentanil | Tramadol + Metoprolol
Number analyzed (Participants) | 44 | 44
minutes | 8.3 (2.1) | 13.4 (4.2)
Statistical Analysis 1: Comparison: Remifentanil vs Tramadol + Metoprolol; Test type: Superiority; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Bleeding Rate
Description: In the end of each surgery, bleeding rate will be calculated as ml/min by dividing total bleeding (amount of blood in the graded suction and sponges minus total irrigation fluid) to the duration of surgery (excluding local anesthetic infiltration, and nasal packing).
Time Frame: throughout surgery, up to 3 hours
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Remifentanil | Tramadol + Metoprolol
Number analyzed (Participants) | 44 | 44
ml/min | 0.53 (0.2) | 0.45 (0.15)
Statistical Analysis 1: Comparison: Remifentanil vs Tramadol + Metoprolol; Test type: Superiority; p = 0.052, t-test, 2 sided

4. Secondary Outcome: Postoperative Pain
Description: Postoperative pain scores on the day of surgery will be evaluated with a visual analog scale (0: no pain, 10: worst pain ever) at the post anaesthetic care unit (PACU), and the surgical ward. The evaluation will begin after the patient arrives at the post anaesthetic care unit, and will continue for 24 hours.
Time Frame: following extubation, up to 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Remifentanil | Tramadol + Metoprolol
Number analyzed (Participants) | 44 | 44
units on a scale
  VAS at arrival to PACU | 3 [2 to 6] | 3 [2 to 3]
  VAS at discharge from PACU | 4 [3 to 5] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Remifentanil vs Tramadol + Metoprolol; Null hypothesis was that the visual analog pain scores (VAS) of patients at arrrival to post anesthetic care unit (PACU) were similar; Test type: Superiority; p = 0.05, Chi-squared
Statistical Analysis 2: Comparison: Remifentanil vs Tramadol + Metoprolol; Null hypothesis was that the visual analog pain scores (VAS) of patients at discharge from post anesthetic care unit (PACU) were similar; Test type: Superiority; p = 0.55, Chi-squared

5. Secondary Outcome: Number of Participants With Postoperative Nausea and Vomiting
Description: Postoperative nausea, retching, and vomiting on the day of surgery will be evaluated with a four-point ordinal scale (0-none, 1-nausea, 2-retching, 3-vomiting) at the post anaesthetic care unit, and the surgical ward. The evaluation will begin after the patient arrives at the post anaesthetic care unit, and will continue for 24 hours.
Time Frame: following extubation, up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Remifentanil | Tramadol + Metoprolol
Number analyzed (Participants) | 44 | 44
Participants | 14 | 10
Statistical Analysis 1: Comparison: Remifentanil vs Tramadol + Metoprolol; Test type: Superiority; p = 0.47, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event data were collected during the whole study period.
Arm/Group | Remifentanil | Tramadol + Metoprolol
Serious Adverse Events (participants affected / at risk) | 21/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remifentanil (N=44) | Tramadol + Metoprolol (N=44)
Intraoperative hypotension (Cardiac disorders) | 3 (8) | 0 (0) — Occurrence of intraoperative hypotension defined as a drop in mean blood pressure by > 30% from baseline.
Intraoperative bradycardia (Cardiac disorders) | 18 (44) | 0 (0) — Occurrence of intraoperative bradycardia defined as heart rate below 50 beats per min.
Intraoperative bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) — Occurrence of intraoperative bleeding serious enough to cause a postponement or cancellation of surgery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remifentanil (N=44) | Tramadol + Metoprolol (N=44)
Adverse hemodynamic event in the surgical ward (Cardiac disorders) | 0 (0) | 0 (0) — Occurrence of any adverse hemodynamic event (hypertensive episode, hypotensive episode, tachycardia, bradycardia).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes